CLINICAL TRIAL: NCT05655247
Title: Partial-thickness/Non-advanced vs. Full-thickness/MCAT Tunnelling for the Treatment of Multiple Gingival Recessions: a Multi-centre Randomized Clinical Trial
Brief Title: Partial-thickness/Non-advanced vs. Full-thickness/MCAT Tunnelling for the Treatment of Multiple Gingival Recessions
Acronym: Tun_RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Principal Investigator, Mario Romandini, Dr., Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MR_03
Record Dates: First submitted 2022-11-29; First posted 2022-12-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split-thickness non-advanced tunnel (Zabalegui et al. 1999) (Experimental)
  Interventions: Procedure: Split-thickness non-advanced tunnel (Zabalegui et al. 1999)
- Full-thickness coronally-advanced tunnel (Aroca et al. 2010) (Active Comparator): Modified Coronally Advanced Tunnel (MCAT)
  Interventions: Procedure: Full-thickness coronally-advanced tunnel (Aroca et al. 2010)

INTERVENTIONS:
Procedure: Split-thickness non-advanced tunnel (Zabalegui et al. 1999) — A split-thickness non-advanced tunnel will be performed according to Zabalegui et al. (1999).
  Arms: Split-thickness non-advanced tunnel (Zabalegui et al. 1999)
Procedure: Full-thickness coronally-advanced tunnel (Aroca et al. 2010) — A full-thickness coronally-advanced tunnel (Modified Coronally Advanced Tunnel - MCAT) will be performed according to Aroca et al. (2010).
  Arms: Full-thickness coronally-advanced tunnel (Aroca et al. 2010)

SUMMARY:
Included patients will be randomly allocated to the test (split-thickness non-advanced tunnel - Zabalegui et al. 1999) or to the control group (full-thickness coronally-advanced tunnel - MCAT - Aroca et al. 2010).

DETAILED DESCRIPTION:
Design: Randomized, clinical, outcome-assessor blinded, multi-centric, superiority trial with two parallel groups and a 1:1 allocation ratio. The follow-up of individual patients will be 6 months (to be extended to 3/5 years if funding will be available)

Patients with a minimum of two-adjacent teeth with RT1 and/or RT2 gingival recessions (at least one with a depth >2 mm) with indication for root coverage treatment will be included. RT2 gingival recessions will be considered not eligible when associated with interproximal exposure of the CEJ.

Mean root coverage (linear) at 6-months will be evaluated as the primary outcome by a blinded outcome assessor.

ELIGIBILITY:
Any patient having a minimum of two adjacent teeth with RT1 and/or RT2 gingival recessions (at least one with a depth >2 mm) with indication for root coverage treatment, being at least 18 years old and able and agreeing to sign a written informed consent form will be potentially eligible for this trial. RT2 gingival recessions will be considered not eligible when associated with interproximal exposure of the CEJ (interdental gingival recession).

In case of multiple RT1/RT2 recessions involving 2 or 3 teeth, at least 2 or 1 more non-included adjacent teeth should respectively be present in order to guarantee a minimum of 4 adjacent teeth (including the included ones) in the region of interest (ROI) for digital scanning.

Patients fitting to all the inclusion criteria as above will be not included in the study if they appear to be unable to attend to the study-related procedures (including the follow-up visits) or if one or more of the following systemic or local exclusion criteria are found in the enrollment phase.

Systemic primary exclusion criteria:

* Compromised general health which contraindicates the study procedures (ASA IV-VI patients);
* Systemic diseases/medications which could influence the outcome of the therapy (e.g., uncontrolled diabetes mellitus);
* Current smokers (self-reported, any type of smoking), users of chewing tobacco, and drug/alcohol abusers;
* Pregnant or nursing women;

Local primary exclusion criteria:

* History of previous periodontal surgery (mucogingival or other) on the teeth to be included;
* Patients having had surgical soft tissue augmentation procedures in the ROI within the previous 12 months;
* Furcation involvement in the teeth to be included;
* Presence of severe tooth malposition, rotation or clinically significant super-eruption in the teeth to be treated;
* Presence of fixed or removable prosthesis in the area to be treated;
* Presence of RT3 gingival recessions in the same surgical area of the treatment.

Secondary exclusion criteria (after initial therapy is provided):

* Not able to achieve good oral hygiene and control gingivitis in the whole of the dentition (FMPS < 20% and FMBS < 20%);
* Persistence of uncorrected gingival trauma from toothbrushing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean Root Coverage (MRC) (6 months) | 6 months after surgery
  Defined as the percentage of root coverage in the mid-buccal aspect obtained with respect to baseline. The MRC will be measured as a percentage (% mm, with probe) 6 months after surgery. Considering the study will also include RT2 gingival recessions (we expect CRC not possible in some cases), the linear 6 months MRC will be evaluated as the primary outcome of the study.

SECONDARY OUTCOMES:
Mean Root Coverage (MRC) (3 months) | 3 months after surgery
  Defined as the percentage of root coverage in the mid-buccal aspect obtained with respect to baseline. The MRC will be measured as a percentage (% mm, with probe) 3 months after surgery.
Complete Root Coverage (CRC) | 3 and 6 months after surgery
  Defined as the presence/absence of complete root coverage in the mid-buccal aspect. It will be measured at 3- and 6-months after surgery and evaluated as linear mid-buccal measurement (mm, with probe).
Recession Reduction (RR) | 3 and 6 months after surgery
  Defined as the reduction in recession in the mid-buccal aspect with respect to baseline. It will be calculated at 3- and 6-months after surgery and evaluated as linear mid-buccal measurement (mm, with probe).
Contact-point/Papilla-tip (DCP) distance changes | 3 and 6 months after surgery
  Defined as the change in the linear distance between the contact point and the top of papilla at the mesial aspect of each tooth (Aroca et al. 2010) with respect to baseline. It will be measured at 3- and 6-months after surgery and evaluated as linear measurement (mm, with probe).
Keratinized Tissue Height (KTH) changes | 3 and 6 months after surgery
  Defined as the linear changes in mid-buccal keratinized tissue height (distance from the gingival margin and the mucogingival junction) with respect to baseline. It will be calculated at 3- and 6-months after surgery and evaluated as linear mid-buccal measurement (mm, with probe).
Probing Pocket Depth (PPD) changes | 3 and 6 months after surgery
  Defined as the changes in PPD (distance from the gingival margin to the bottom of the probeable sulcus) with respect to baseline. It will be calculated at 3- and 6-months after surgery and evaluated only as linear mid-buccal measurement (mm, with probe).
Clinical Attachment Level (CAL) changes | 3 and 6 months after surgery
  Defined as the changes in CAL (distance from the CEJ to the bottom of the probeable sulcus) with respect to baseline. It will be calculated at 3- and 6-months after surgery and evaluated only as linear mid-buccal measurement (mm, with probe).
Dental hypersensitivity (DH) | 3 and 6 months after surgery
  Assessed by 10 s air spray applied to the buccal cervical area. It will be evaluated at baseline and at 3- and 6-months after surgery.
Root-coverage Esthetic Score (RES) | 3 and 6 months after surgery
  Evaluated at 3- and 6-months according to Cairo et al. (2009).
Digital Mean Root Coverage (dMRC) | 3 and 6 months after surgery
  Defined as the percentage of root surface coverage obtained with respect to baseline. The sMRC will be measured at 3- and 6-months after surgery. It will be assessed as buccal surface measurement (% mm2, digital assessment).
Digital Complete Root Coverage (dCRC) | 3 and 6 months after surgery
  Defined as the presence/absence of complete root surface coverage. It will be measured at 3- and 6-months after surgery and evaluated as buccal surface measurement (mm2, digital assessment).
Digital Recession Reduction (dRR) | 3 and 6 months after surgery
  Defined as the reduction in recession surface with respect to baseline. It will be calculated at 3- and 6-months after surgery and evaluated as buccal surface measurement (mm2, digital assessment).
Digital Contact-point/Papilla-tip (dDCP) distance changes | 3 and 6 months after surgery
  Defined as the changes in the area between the contact point and the top of papilla at the mesial aspect of each tooth with respect to baseline. It will be measured at 3- and 6-months after surgery and evaluated as area measurement (mm2, digital assessment).
Digital Gingival thickness (dGT) | 3 and 6 months after surgery
  It will be measured both at the gingival margin and 1-mm apically. It will be assessed as a mid-buccal thickness measurement (mm, digital assessment) at 3- and 6-months after surgery.
Digital Keratinized Tissue Height (dKTH) changes | 3 and 6 months after surgery
  Defined as the changes in keratinized tissue surface (surface delimited apico-coronally by the gingival margin and the mucogingival junction and mesio-distally by the projection of a line passing by the contact-point and perpendicular to the occlusal aspect of each tooth) with respect to baseline. It will be calculated at 3- and 6-months after surgery and evaluated as buccal surface measurement (mm2, digital assessment).

OTHER OUTCOMES:
PROMs - Pain | Just after surgery, 12 hours and 1, 2, 3, 4, 5, 6, 7, 14 days after surgery
  The patient will self-report on a 100-mm VAS scale ranging from 0 (no pain whatsoever) to 100 (worst pain imaginable) the perceived pain. The pain will be reported just after surgery, 12 hours post-operatively and 1, 2, 3, 4, 5, 6, 7, 14 days post-operatively in the evening, preferably at the same time.
PROMs - Time to non-significant pain | 14 days after surgery
  It will be defined as the time (days) to reach a pain VAS<10.
PROMs - Number of analgesic tablets | 14 days after surgery
  The patient will document in the evening, preferably at the same time, the number of ibuprofen tablets taken each day from day-0 to day-7 and at day-14 post-surgery.
PROMs - Swelling | Just after surgery, 12 hours and 1, 2, 3, 4, 5, 6, 7, 14 days after surgery
  The patient will self-report on a 100-mm VAS scale ranging from 0 (no swelling whatsoever) to 100 (worst swelling imaginable) the perceived swelling. The swelling will be reported just after surgery, 12 hours post-operatively and 1, 2, 3, 4, 5, 6, 7, 14 days post-operatively in the evening, preferably at the same time.
PROMs - Bleeding | Just after surgery, 12 hours and 1, 2, 3, 4, 5, 6, 7, 14 days after surgery
  The patient will self-report on a 100-mm VAS scale ranging from 0 (no bleeding whatsoever) to 100 (continuous copious bleeding) the perceived bleeding. The bleeding will be reported just after surgery, 12 hours post-operatively and 1, 2, 3, 4, 5, 6, 7, 14 days post-operatively in the evening, preferably at the same time.
PROMs - Discomfort during surgery | Just after surgery
  The patient will answer on a 100-mm VAS scale just after the surgery to the following question: "How did you perceive the procedure?" (Burkhardt et al. 2015). The VAS scale will range from 0 (no problem whatsoever) to 100 (unbearable).
PROMs - Aesthetic consequences (self-evaluation) | 6 months after surgery
  The patient will self-report on a 100-mm VAS scale ranging from 0 (terrible) to 100 (perfect) the perceived aesthetic of the included zone. The aesthetic self-evaluation will be completed 6 months post-surgery.
PROMs - Satisfaction (self-evaluation) | 6 months after surgery
  The patient will self-report on a 100-mm VAS scale ranging from 0 (terrible) to 100 (perfect) the overall satisfaction for the treatment of the included zone. The satisfaction self-evaluation will be completed at 6-months post-surgery.
PROMs - Oral Health Impact Profile-14 (OHIP-14) | 1, 2, 3, 4, 5, 6, 7, 14 days, as well as 6 months, after surgery
  The OHIP-14 questionnaire will be evaluated at 1, 2, 3, 4, 5, 6, 7, 14 days and 6 months post-surgery.
PROMs - Patient concerns with gingival recession | 6 months after surgery
  Patient concerns with gingival recession will be assessed with a condition-specific health-related quality-of-life instrument (Tonetti et al. 2018) assessing the level of concern in terms of aesthetics, sensitivity to cold, sensitivity to brushing, root/tooth wear, development of cavity and fear to lose the involved teeth using a questionnaire on a 5-point Likert scale at 6 months.
Duration of surgery | During surgery
  The time in minutes of the net (excluding time used for photographs or other non-surgery related things) duration of the surgery in the recipient site (after palate suture), from the first incision to the completion of the last suture (the composite stops placement in the control group will be considered within the duration of surgery).
Early Wound Healing | 1 and 2 weeks after surgery
  It will be evaluated by the outcome assessor on a 100-mm VAS scale ranging from 0 (very bad) to 100 (very good). The early wound healing will be evaluated at 1 and 2 weeks post-surgery.
Micro-vascularization (eco-doppler) | Just after surgery; 1, 2, 4 weeks after surgery; 3 and 6 months after surgery
  It will be evaluated on patients treated in one of the centers, using a 3D printed stent, just after surgery, and at 1-, 2- and 4-week, as well as 3- and 6-months examinations, after-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Taranto, Italy

REFERENCES:
- [Background] Aroca S, Keglevich T, Nikolidakis D, Gera I, Nagy K, Azzi R, Etienne D. Treatment of class III multiple gingival recessions: a randomized-clinical trial. J Clin Periodontol. 2010 Jan;37(1):88-97. doi: 10.1111/j.1600-051X.2009.01492.x. Epub 2009 Nov 30. PMID 19968743
- [Background] Zabalegui I, Sicilia A, Cambra J, Gil J, Sanz M. Treatment of multiple adjacent gingival recessions with the tunnel subepithelial connective tissue graft: a clinical report. Int J Periodontics Restorative Dent. 1999 Apr;19(2):199-206. PMID 10635186